CLINICAL TRIAL: NCT07155122
Title: Efficacy and Safety of Serplulimab Combined With Etoposide and Cisplatin as Neoadjuvant Therapy in Limited-Stage Small-Cell Carcinoma of the Esophageal : A Single-Arm, Phase II Clinical Study
Brief Title: Efficacy and Safety of Serplulimab Combined With Etoposide and Cisplatin as Neoadjuvant Therapy in Limited-Stage Small-Cell Carcinoma of the Esophageal
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFWM-01
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Small-Cell Carcinoma of the Esophageal
Keywords: Small Cell Carcinoma of the Esophagus; Neoadjuvant Therapy; Serplulimab
MeSH Terms: interventions — Etoposide; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serplulimab Combined With Etoposide and Cisplatin (Experimental)
  Interventions: Drug: Drug: Serplulimab; Drug: Drug: Etoposide; Drug: Drug: Chemotherapy

INTERVENTIONS:
Drug: Drug: Serplulimab — serplulimab Serplulimab , 300mg, D1, intravenous drip , Q3W.
Drug: Drug: Etoposide — Etoposide, 60-100 mg/m², D1-3 or D1-5, intravenous drip, Q3W
Drug: Drug: Chemotherapy — Cisplatin, 50-75 mg/m², D2, intravenous drip, Q3W. Or Carboplatin, AUC 5, D2, intravenous drip, Q3W.

SUMMARY:
This study is a prospective, single-center, single-arm phase II clinical trial designed to evaluate the efficacy and safety of serplulimab in combination with etoposide and platinum-based chemotherapy as neoadjuvant treatment for patients with limited-stage small cell carcinoma of the esophagus (SCCE). The primary endpoint is the pathological complete response (pCR) rate. Secondary endpoints include major pathological response (MPR) rate, objective response rate (ORR), disease control rate (DCR), disease-free survival (DFS), overall survival (OS) and safety. A total of 15 patients are expected to be enrolled.

DETAILED DESCRIPTION:
Small cell carcinoma of the esophagus (SCCE) is a rare but highly aggressive subtype of esophageal cancer, accounting for approximately 0.4% to 2.8% of all esophageal malignancies. It is characterized by high malignancy, a strong tendency for early metastasis, and poor prognosis. Currently, there is no standardized treatment regimen for SCCE. The efficacy of chemotherapy is limited, and resistance often develops rapidly. With the advancement of cancer immunotherapy, PD-1/PD-L1 inhibitors have demonstrated significant efficacy across various solid tumors. Given the biological and molecular similarities between SCCE and small cell lung cancer (SCLC), immune checkpoint inhibitors may offer a novel therapeutic avenue for patients with SCCE.This study is a prospective, single-center, single-arm phase II clinical trial designed to evaluate the efficacy and safety of serplulimab in combination with etoposide and platinum-based chemotherapy as neoadjuvant treatment for patients with limited-stage small cell carcinoma of the esophagus (SCCE). The preoperative neoadjuvant treatment drugs are f serplulimab + etoposide + platinum, with a cycle of 3 weeks. The combined treatment is given for 2 cycles. Radical resection of esophageal cancer is performed 4 to 6 weeks after the last dose. After surgery, the researcher decides whether to continue adjuvant treatment based on the pathological condition.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥18 years;
2. Histologically or cytologically confirmed diagnosis of SCCE prior to initiation of any treatment;
3. Clinical stage cT2-4aNxM0 or cT1N+M0, corresponding to limited-stage SCCE based on the American Joint Committee on Cancer (AJCC) staging systemand the Veterans Administration Lung Study Group (VALSG) classification for small cell lung cancer;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. For women of childbearing potential, a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent) within 48 hours prior to the first administration of the study drug. Female patients must not be breastfeeding;
6. All participants were required to undergo baseline laboratory evaluations within two weeks prior to treatment, and the results must meet the following criteria (based on CTCAE version 5.0):White blood cell count ≥ 3,000/μL; Absolute neutrophil count ≥ 1,500/μL; Platelet count ≥ 75 × 10³/μL; Hemoglobin ≥ 9.0 g/dL; Creatinine clearance > 30 mL/min (calculated by the Cockcroft-Gault formula); Aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤ 3 × ULN; Total bilirubin ≤ 1.5 × ULN.
7. Written informed consent must be obtained prior to the initiation of any study-related procedures. The informed consent form must be reviewed and approved by the institutional ethics committee. Participants must be willing and able to comply with the study protocol, including treatment, visit schedule, biospecimen collection, and other study-related requirements.

Exclusion Criteria:

1. Patients with esophageal cancer of any histological type other than small cell carcinoma;
2. Patients clinically staged as cT4bNanyM0, cTanyN3M0, or cTanyNanyM1;
3. History of other malignancies, unless the patient has achieved complete remission for at least 3 years prior to enrollment and does not require or is not expected to require additional treatment during the study period;
4. Known or suspected active autoimmune diseases. However, patients with type I diabetes mellitus, hypothyroidism requiring only hormone replacement therapy, skin disorders not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger may be included;
5. Systemic treatment with corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days prior to administration of study drugs. Inhaled, topical, or adrenal replacement corticosteroids at doses >10 mg/day of prednisone equivalent are permitted in the absence of active autoimmune disease;
6. Prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibodies, or any other agents targeting T-cell co-stimulatory or immune checkpoint pathways;
7. Any serious or uncontrolled medical conditions or active infections that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, or may interfere with the patient's ability to receive the planned treatment;
8. Known history of HIV infection or acquired immunodeficiency syndrome (AIDS). (Note: HIV testing must be performed at study centers where required by local regulations);
9. Clinically significant arrhythmias, myocardial ischemia, severe atrioventricular block, heart failure, or significant valvular heart disease; severe pulmonary dysfunction; hematologic, hepatic, or renal dysfunction precluding tolerance to chemoradiotherapy; severe bone marrow failure; or uncontrolled infections;
10. Inability to comply with the study protocol and procedures;
11. Known hypersensitivity to any component of the investigational agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate (pCR) | Each 2 cycles (each cycle is 21 days).

SECONDARY OUTCOMES:
Major pathological response rate (MPR) | Each 2 cycles (each cycle is 21 days).
Objective response rate (ORR) | Each 2 cycles (each cycle is 21 days).
Disease control rate (DCR) | Each 2 cycles (each cycle is 21 days).
Disease-free survival (DFS) | 36-months
Overall survival (OS) | 36-months
Safety: The incidence and severity of adverse events (AE) and serious adverse events (SAE) | From the time the subject is enrolled until the 90th day after the last dose